CLINICAL TRIAL: NCT02683174
Title: Diagnostic Yield of an Ambulatory Patch Monitor in Emergency Department Syncope Patients Unexplained After Emergency Department Evaluation: A Pilot Study (PATCH-ED)
Brief Title: Diagnostic Yield of an Ambulatory Patch Monitor in Unexplained Emergency Department Syncope: A Pilot Study (PATCH-ED)
Acronym: PATCH-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015/0225; 179127 (Other Grant/Funding Number: IRAS project ID); 19511 (Other: UKCRN portfolio ID)
Record Dates: First submitted 2016-02-05; First posted 2016-02-17 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2016-09

CONDITIONS: Syncope
Keywords: syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single study arm (Experimental): All enrolled patients will be fitted with a novel ambulatory patch (ZIO®Patch), which continuously records heartbeats for up to 14 days. Brain natriuretic peptide (BNP) and hs-troponin I at 0 and 3 hours post ED attendance
  Interventions: Device: Novel ambulatory patch (ZIO® XT Patch); Biological: BNP and hs-troponin I at 0 and 3 hours post ED attendance

INTERVENTIONS:
Device: Novel ambulatory patch (ZIO® XT Patch) — All enrolled patients will be fitted with a novel ambulatory patch (ZIO® XT Patch)
Biological: BNP and hs-troponin I at 0 and 3 hours post ED attendance — All patients will have quantification of hs-troponin I (ARCHITECTSTAT high-sensitivity troponin I assay) and BNP (ALERE TRIAGE point-of-care BNP test; ALERE, San Diego, USA; www.alere.co.uk) at 0 and 3 hours post ED attendance.

SUMMARY:
Syncope is a common Emergency Department (ED) presentation but the underlying diagnosis is not apparent in 60% of patients after assessment and serious adverse event rate is 7% at one month with most having acute cardiovascular events, also more likely to be unexplained after ED assessment. Many cardiovascular events are due to arrhythmia, difficult for clinicians to diagnose, as examination and Electrocardiogram (ECG) findings may both be normal and symptoms have resolved by the time the patient gets to the ED. Currently establishing a cardiac arrhythmia as the cause of syncope rests on correlating the arrhythmia with symptoms using monitoring devices such as Holter but these all have significant drawbacks. The clinical challenge in the ED is therefore to identify the moderate and high-risk patients and refer them for further investigation and monitoring if appropriate. The logistics of arranging follow up within a timely period of the patient's ED visit is often problematic for a variety of reasons including availability of timely specialty outpatient appointments, a lack of consensus of the specialty to whom the syncope patient should be referred (cardiology, medicine, neurology, general practice) and availability of Holter and other monitoring devices. For this reason most high and medium risk patients are admitted to hospital.

Previous syncope clinical decision rules have not been well adopted due to their lack of sensitivity and specificity probably due to the varied and heterogeneous nature of potentially serious causes. However, the majority of patients with syncope have no serious underlying pathology and do not require hospitalisation. Rather than continued attempts at risk stratification of outcome based on presentation, more research is required into how we can better improve diagnosis and therefore treatment in order to provide improved patient benefit. We believe that ambulatory patch monitoring will allow better and earlier arrhythmia detection and plan to assess the ability of a 14-day ambulatory patch to detect serious arrhythmic outcomes at 90 days.

DETAILED DESCRIPTION:
There are around 650,000 ED syncope presentations a year in the United Kingdom (UK). Serious underlying conditions can present with syncope and one-month serious adverse outcome is around 7% with 50% being cardiovascular. The treating ED clinician is not always able to rule out serious pathology as the patient is commonly fully recovered on arrival in the ED, despite the underlying cause being potentially life threatening should it recur again. Whilst most patients do not have a serious underlying cause and therefore do not require hospitalisation, the concern of the ED clinician about missing a serious underlying cause (especially cardiovascular ones) means that 50% of syncope patients are admitted to hospital.

Despite research identifying high-risk demographic, historical and examination variables, clinical decision rules have not been well adopted due to their lack of sensitivity and specificity probably due to the varied and heterogeneous nature of potentially serious causes. Rather than continued attempts at risk stratification of outcome based on presentation, more research is required into how we can better improve diagnosis and therefore treatment in order to provide improved patient benefit.

Cardiovascular causes of syncope fall into two main categories, arrhythmia (e.g. ventricular tachycardia (VT), 2nd degree Mobitz II, 3rd degree atrioventricular block or symptomatic bradycardia) and structural (e.g. aortic stenosis). It is arrhythmia that is most difficult for the ED clinician to diagnose in the ED as examination and presenting Electrocardiogram ECG may both be normal. It is for this reason that arrhythmia makes up a large number of subsequent serious outcomes in syncope patients whose syncopal cause is unexplained after ED assessment.

The current main method for establishing a cardiac arrhythmia as the cause of syncope rests on the correlation of the arrhythmia with symptoms (which will have resolved by the time the patient gets to the ED). The clinical challenge in the ED is therefore to identify the moderate and high-risk patients and refer them for further investigation and monitoring if appropriate. The logistics of arranging follow up within a timely period of the patient's ED visit is often problematic for a variety of reasons including availability of timely specialty outpatient appointments, a lack of consensus of the specialty to whom the syncope patient should be referred (cardiology, medicine, neurology, general practice) and availability of Holter and other monitoring devices. For this reason most high and medium risk patients are admitted to hospital.

The investigation of cardiac arrhythmias is usually initiated with the Holter monitor which uses a continuous recording over a 24 or 48-hour period. The Holter allows detection of baseline rhythm, arrhythmia and conduction abnormalities. Holters however are bulky and inconvenient for the patient to wear, the transmission of data is not patient dependent and non-compliance with both device use and maintaining a written symptom log, limits its diagnostic utility. The lack of extended monitoring reduces diagnostic yield to typically less than 20%. Bass reported a diagnostic yield of 15% with 24-hour Holter monitoring that did not increase even if the device was applied for 72 hours.

For these reasons, the use of Holter monitors is not universal in medium and high-risk syncope patients. In one UK ED study, only 158 of 540 (29%) admitted syncope patients underwent 24 hour monitoring (which in the majority comprised ward telemetry rather than Holter). There are other devices available to the Cardiologist to investigate syncope patients who are classified as European Society of Cardiology (ESC) medium and high-risk and whose Holter investigation is unrevealing. Event recorders do not record a continuous ECG but require patient activation at the time of symptoms and must be applied to the chest wall at the time of the event and must be activated by the patient. A brief, typically 90-second, single lead ECG recording is captured and stored. Because of limited data storage capability, data must be transmitted to a monitoring centre for validation and analysis. Event recorders can be used for cardiac monitoring over longer periods of time but the big drawback is that they must be activated following symptom onset, which may be difficult to achieve if the patient has suffered syncope or an injury related to the event. Finally, these devices cannot be used to document asymptomatic arrhythmias.

External continuous loop recorders are attached to the patient by chest electrodes or a wristband. They continuously record the ECG but only save data if activated by the patient. The continuous looping memory feature allows the device to store a fixed length of pre-activation and post-event ECG data. Mobile cardiac telemetry systems provide up to 30 days of real-time continuous cardiac monitoring without the need for patient activation or data transmission. These devices are expensive, require electrodes and bulky recording devices, and produce a large amount of data, which requires sifting. Implantable loop recorders are surgically implanted subcutaneous devices that continuously record single-lead ECG signal through 2 electrodes. They are very expensive and necessitate an invasive surgical procedure. For patients admitted to hospital and who are placed on telemetry, there is also lack of consensus on the optimal duration of monitoring. Typically higher risk patients are monitored for 24 hours and discharged without a diagnosis if their ECG tracing has been uneventful during this time period.

In order to solve these problems, a novel ambulatory cardiac monitoring device that can easily be applied to ED patients has recently been developed. The ZIO®XT Patch (iRhythm Technologies, Inc. San Francisco, California; http://www.irhythmtech.com/zio-services.php) is non-invasive, water-resistant, has no leads or wires, is discrete to wear and has been approved for clinical use in the UK. It continuously monitors the heart for up to 14 days including during sleep, in the shower, and during moderate exercise and has a large button on top for patients to capture symptomatic events. When patients reach the end of their monitoring period, they simply mail the device back to the company where analysis is undertaken.

The ZIO®XT Patch is well tolerated for prolonged monitoring and compliance is excellent with studies demonstrating a mean monitoring wear time of 10.8 days (range 4-14 days) and 10.9 days (median 13.0 days). Barrett et al showed that 80% of patients who had worn a Holter monitor for 24 hours, and a ZIO®XT Patch for up to 14 days, preferred the ZIO Patch. Single channel ECG data quality is also excellent with one study showing more than 98% of the total recording time was analysable, and a second study showing a median analysable time of 99% of the total wear time. Compliance with returning the device is also good. In a study of 174 ED with indications for monitoring (syncope, dizziness and palpitations), all patients mailed back their devices.

Several studies have shown that ZIO®XT Patch has a higher diagnostic yield for arrhythmias than traditional 24-48 hour Holter monitoring and importantly can also efficiently characterise symptomatic patients without significant arrhythmia. The absence of an arrhythmia during syncope, palpitations or a triggered event does not by itself provide a definitive diagnosis but does allow the clinician to exclude an arrhythmia as a potential cause and is thus clinically useful. Over half of patients (53.4%) in one study did not have an arrhythmia despite a triggered event. This allows the clinician to potentially exclude an arrhythmia as an etiology of the patient's symptoms and potentially avoid further cardiac evaluation.

Camm et al showed in a study on patients with arrhythmogenic right ventricular dysplasia (ARVD), that over the total wear time of both devices, the ZIO®XT Patch detected more premature ventricular contraction events than a 24 hour Holter monitor. Barrett et al showed ZIO®XT Patch had a 57% greater diagnostic yield than a 24 hour Holter monitor, and Schreiber at al demonstrated an overall diagnostic yield of 63% in ED patients with indications for monitoring. This study also showed that 48% of patients had ≥1 arrhythmia and 10% were symptomatic at the time of their arrhythmia. Median time to first arrhythmia was 1.0 days (IQR 0.2-2.8) and median time to first symptomatic arrhythmia was 1.5 days (IQR 0.4-6.7). 54% of symptomatic patients did not have any arrhythmia during their triggered events.

In a study looking at ZIO®XT Patch use in outpatients with clinical indications for monitoring (15% of whom had syncope), of the 60% of patients who had an arrhythmia detected, 30% had their first arrhythmia and 51% had their first symptom-triggered arrhythmia occur after the initial 48-hour period. Mean time to first arrhythmia was 1.7 days (median 0.8) and mean time to first symptomatic arrhythmia was 3.0 days (median 2.1).

This novel ambulatory cardiac monitoring device should allow much earlier arrhythmia detection in more patients allowing better diagnosis and subsequent treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 years or over presenting within 6 hours of an episode of syncope and whose syncope remains unexplained after ED assessment. Syncope will be defined as a transient loss of consciousness (TLOC) with inability to maintain postural tone and immediate complete spontaneous recovery without medical intervention (to preexisting mental status and neurologic function)

Exclusion Criteria:

* Obvious underlying cause after ED assessment,
* Alcohol or illicit drugs as presumptive cause of TLOC [24],
* Epileptic seizure as presumptive cause of TLOC (seizure activity with a >15 min witness reported post-ictal phase) [24],
* Stroke ⁄ transient ischemic attack as presumptive cause of TLOC [24],
* Head trauma followed by TLOC [24],
* Hypoglycemia as presumptive cause of TLOC [24],
* No consent i.e. patient lacking capacity,
* Previous recruitment into the study,
* Patient in custody or prison.

Obvious underlying causes will be defined as:

* Clinical history of vasovagal syncope i.e. pre-syncope symptoms and low-risk patient according to current ESC guidelines [14],
* Arrhythmia on ED ECG thought to have caused syncope,
* Arrhythmia on pre-hospital ECG causing syncope,
* Pulmonary embolism (PE) diagnosed on Computed Tomography Pulmonary Angiography (CTPA; or equivalent e.g. symptoms of PE plus positive leg ultrasound scan/ventilation-perfusion scan/echo),
* Postural hypotension (postural drop >20 mmHg in ED with symptoms during test and suggestive history),
* Myocardial Infarction [25],
* CT brain or clinical signs/symptoms in ED showing cerebrovascular accident or subarachnoid haemorrhage,
* Evidence of haemorrhage in ED thought to have caused syncope,
* Other obvious cause of syncope apparent in ED.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-11-01; Primary Completion 2017-06-13 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Reed, MA FCEM MD, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be available from 6 months after final publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available from 6 months after final publication with no end date.
Access Criteria: Please contact CI

REFERENCES:
- [Background] Reed MJ, Newby DE, Coull AJ, Prescott RJ, Jacques KG, Gray AJ. The ROSE (risk stratification of syncope in the emergency department) study. J Am Coll Cardiol. 2010 Feb 23;55(8):713-21. doi: 10.1016/j.jacc.2009.09.049. PMID 20170806
- [Background] Reed MJ, Henderson SS, Newby DE, Gray AJ. One-year prognosis after syncope and the failure of the ROSE decision instrument to predict one-year adverse events. Ann Emerg Med. 2011 Sep;58(3):250-6. doi: 10.1016/j.annemergmed.2010.12.021. Epub 2011 Feb 2. PMID 21288597
- [Background] Martin TP, Hanusa BH, Kapoor WN. Risk stratification of patients with syncope. Ann Emerg Med. 1997 Apr;29(4):459-66. doi: 10.1016/s0196-0644(97)70217-8. PMID 9095005
- [Background] Oh JH, Hanusa BH, Kapoor WN. Do symptoms predict cardiac arrhythmias and mortality in patients with syncope? Arch Intern Med. 1999 Feb 22;159(4):375-80. doi: 10.1001/archinte.159.4.375. PMID 10030311
- [Background] Colivicchi F, Ammirati F, Melina D, Guido V, Imperoli G, Santini M; OESIL (Osservatorio Epidemiologico sulla Sincope nel Lazio) Study Investigators. Development and prospective validation of a risk stratification system for patients with syncope in the emergency department: the OESIL risk score. Eur Heart J. 2003 May;24(9):811-9. doi: 10.1016/s0195-668x(02)00827-8. PMID 12727148
- [Background] Sarasin FP, Hanusa BH, Perneger T, Louis-Simonet M, Rajeswaran A, Kapoor WN. A risk score to predict arrhythmias in patients with unexplained syncope. Acad Emerg Med. 2003 Dec;10(12):1312-7. doi: 10.1111/j.1553-2712.2003.tb00003.x. PMID 14644781
- [Background] Quinn JV, Stiell IG, McDermott DA, Sellers KL, Kohn MA, Wells GA. Derivation of the San Francisco Syncope Rule to predict patients with short-term serious outcomes. Ann Emerg Med. 2004 Feb;43(2):224-32. doi: 10.1016/s0196-0644(03)00823-0. PMID 14747812
- [Background] Quinn J, McDermott D, Stiell I, Kohn M, Wells G. Prospective validation of the San Francisco Syncope Rule to predict patients with serious outcomes. Ann Emerg Med. 2006 May;47(5):448-54. doi: 10.1016/j.annemergmed.2005.11.019. Epub 2006 Jan 18. PMID 16631985
- [Background] Costantino G, Perego F, Dipaola F, Borella M, Galli A, Cantoni G, Dell'Orto S, Dassi S, Filardo N, Duca PG, Montano N, Furlan R; STePS Investigators. Short- and long-term prognosis of syncope, risk factors, and role of hospital admission: results from the STePS (Short-Term Prognosis of Syncope) study. J Am Coll Cardiol. 2008 Jan 22;51(3):276-83. doi: 10.1016/j.jacc.2007.08.059. PMID 18206736
- [Background] Del Rosso A, Ungar A, Maggi R, Giada F, Petix NR, De Santo T, Menozzi C, Brignole M. Clinical predictors of cardiac syncope at initial evaluation in patients referred urgently to a general hospital: the EGSYS score. Heart. 2008 Dec;94(12):1620-6. doi: 10.1136/hrt.2008.143123. Epub 2008 Jun 2. PMID 18519550
- [Background] Cheung CC, Kerr CR, Krahn AD. Comparing 14-day adhesive patch with 24-h Holter monitoring. Future Cardiol. 2014 May;10(3):319-22. doi: 10.2217/fca.14.24. PMID 24976467
- [Background] Bass EB, Curtiss EI, Arena VC, Hanusa BH, Cecchetti A, Karpf M, Kapoor WN. The duration of Holter monitoring in patients with syncope. Is 24 hours enough? Arch Intern Med. 1990 May;150(5):1073-8. PMID 2331188
- [Background] Tattersall LC, Reed MJ. The inpatient management of syncope. Emerg Med J. 2010 Nov;27(11):870-2. doi: 10.1136/emj.2010.092924. Epub 2010 Aug 3. PMID 20682959
- [Background] Task Force for the Diagnosis and Management of Syncope; European Society of Cardiology (ESC); European Heart Rhythm Association (EHRA); Heart Failure Association (HFA); Heart Rhythm Society (HRS); Moya A, Sutton R, Ammirati F, Blanc JJ, Brignole M, Dahm JB, Deharo JC, Gajek J, Gjesdal K, Krahn A, Massin M, Pepi M, Pezawas T, Ruiz Granell R, Sarasin F, Ungar A, van Dijk JG, Walma EP, Wieling W. Guidelines for the diagnosis and management of syncope (version 2009). Eur Heart J. 2009 Nov;30(21):2631-71. doi: 10.1093/eurheartj/ehp298. Epub 2009 Aug 27. No abstract available. PMID 19713422
- [Background] Rosenberg MA, Samuel M, Thosani A, Zimetbaum PJ. Use of a noninvasive continuous monitoring device in the management of atrial fibrillation: a pilot study. Pacing Clin Electrophysiol. 2013 Mar;36(3):328-33. doi: 10.1111/pace.12053. Epub 2012 Dec 13. PMID 23240827
- [Background] Tung CE, Su D, Turakhia MP, Lansberg MG. Diagnostic Yield of Extended Cardiac Patch Monitoring in Patients with Stroke or TIA. Front Neurol. 2015 Jan 12;5:266. doi: 10.3389/fneur.2014.00266. eCollection 2014. PMID 25628595
- [Background] Barrett PM, Komatireddy R, Haaser S, Topol S, Sheard J, Encinas J, Fought AJ, Topol EJ. Comparison of 24-hour Holter monitoring with 14-day novel adhesive patch electrocardiographic monitoring. Am J Med. 2014 Jan;127(1):95.e11-7. doi: 10.1016/j.amjmed.2013.10.003. Epub 2013 Oct 15. PMID 24384108
- [Background] Schreiber D, Sattar A, Drigalla D, Higgins S. Ambulatory cardiac monitoring for discharged emergency department patients with possible cardiac arrhythmias. West J Emerg Med. 2014 Mar;15(2):194-8. doi: 10.5811/westjem.2013.11.18973. PMID 24672611
- [Background] Turakhia MP, Hoang DD, Zimetbaum P, Miller JD, Froelicher VF, Kumar UN, Xu X, Yang F, Heidenreich PA. Diagnostic utility of a novel leadless arrhythmia monitoring device. Am J Cardiol. 2013 Aug 15;112(4):520-4. doi: 10.1016/j.amjcard.2013.04.017. Epub 2013 May 11. PMID 23672988
- [Background] Camm CF, Tichnell C, James CA, Murray B, Porterfield F, Te Riele AS, Tandri H, Calkins H. Premature ventricular contraction variability in arrhythmogenic right ventricular dysplasia/cardiomyopathy. J Cardiovasc Electrophysiol. 2015 Jan;26(1):53-7. doi: 10.1111/jce.12544. Epub 2014 Oct 27. PMID 25215858
- [Derived] Reed MJ, Grubb NR, Lang CC, Gray AJ, Simpson K, MacRaild A, Weir CJ. Diagnostic yield of an ambulatory patch monitor in patients with unexplained syncope after initial evaluation in the emergency department: the PATCH-ED study. Emerg Med J. 2018 Aug;35(8):477-485. doi: 10.1136/emermed-2018-207570. Epub 2018 Jun 19. PMID 29921622

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Study Arm
Started | 86
Completed | 86
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Study Arm
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (19.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Ambulatory Patch Monitor Participants Having Significant Symptomatic Arrhythmia
Description: Significant arrhythmia will be defined as:
  * Non-symptomatic ventricular tachycardia < 30 seconds,
  * Symptomatic sinus bradycardia < 60 beats/minute (but >40 or less than 30 seconds),
  * Asymptomatic sinus bradycardia < 40 beats/minute,
  * Sick sinus syndrome with alternating sinus bradycardia and tachycardia,
  * Sinus pause > 3 seconds (but less than 6 seconds),
  * Symptomatic Mobitz type I atrioventricular heart block,
  * Junctional/idioventricular rhythm,
  * Symptomatic supraventricular tachycardia with rate > 100/minute,
  * Symptomatic atrial flutter/fibrillation with ventricular rate >100/min,
  * Symptomatic atrial flutter/fibrillation with ventricular rate <60/min
  Arrhythmias will also be defined as symptomatic (i.e. concurrent light-headedness/dizziness, syncope/presyncope with arrhythmia) or asymptomatic.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Groups:
- Study Group: Patients 16 years or over presenting within 6 hours of unexplained syncope were fitted in the ED with an ambulatory patch ECG recorder (Zio XT monitor), which continuously records a single-lead ECG for up to 14 days.
Arm/Group | Study Group
Number analyzed (Participants) | 86
Participants | 9

2. Secondary Outcome: Median Time to Detection of Significant Symptomatic Arrhythmia
Description: Median time to detection of significant symptomatic arrhythmia by ambulatory patch monitor
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Study Group
Number analyzed (Participants) | 86
days | 19 [4 to 30]

3. Secondary Outcome: Number of Participants With Arrhythmia
Description: Prevalence of arrhythmia including serious significant arrhythmia, significant arrhythmia and symptomatic arrhythmia in ED syncope patients unexplained after ED evaluation.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Study Arm
Number analyzed (Participants) | 86
Participants
  Yes | 24
  No | 62

4. Secondary Outcome: Number of Participants Who Agreed or Strongly Agreed That the Patch Monitor Was Easy to Use.
Description: Number of participants who agreed or strongly agreed that the patch monitor was easy to use. Patient patch satisfaction (postal questionnaire).
Time Frame: 90 days
Population: All study participants who returned the participant patch satisfaction postal questionnaire (n=47).
Measure: Count of Participants; unit: Participants
Arm/Group | Single Study Arm
Number analyzed (Participants) | 47
Participants
  Yes | 43
  No | 4

5. Secondary Outcome: Median Device Wear Time
Description: Patch compliance described by median device wear time
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Single Study Arm
Number analyzed (Participants) | 86
days | 13.6 [11.8 to 14.0]

6. Secondary Outcome: Number of Participants With Significant Arrhythmia Requiring Referral.
Description: Number of participants with significant underlying arrhythmic pathology on ambulatory patch monitoring requiring referral.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Study Arm
Number analyzed (Participants) | 86
Participants | 12

7. Secondary Outcome: Number of Participants With All Cause Serious Outcome
Description: All cause serious outcome will be a composite of:
  * All cause death,
  * Major adverse cardiac events [MACE]
    * Myocardial infarction [25],
    * Significant arrhythmia [25],
    * Significant Structural Heart Disease [23],
    * Positive Electrophysiology Study Findings [25]
    * Permanent pacemaker or defibrillator placement,
    * Coronary artery bypass graft or coronary artery stent,
    * Cardiac valve surgery,
    * Elective cardioversion in the absence of objective evidence that tachyarrhythmia is responsible for the syncope,
    * Balloon-pump insertion,
    * Heart transplant,
    * Initiation of anti-arrhythmia medical therapy,
    * Ventricular assist device
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Study Arm
Number analyzed (Participants) | 86
Participants | 26

ADVERSE EVENTS:
Time Frame: 90 days
Description: Patients were followed up at 90 days after presentation through hospital and primary care electronic patient record (EPR) systems. Patients who had left the NHS Lothian area after 1 month were contacted by telephone.
Groups:
- Study Arm: All enrolled patients will be fitted with a novel ambulatory patch (ZIO® XT Patch)
Arm/Group | Study Arm
All-Cause Mortality (participants affected / at risk) | 1/86
Serious Adverse Events (participants affected / at risk) | 26/86
Other Adverse Events (participants affected / at risk) | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=86)
Significant arrhythmia (Cardiac disorders) | 24 (24)
Permanent pacemaker or defibrillator placement (Cardiac disorders) | 4 (4)
Coronary artery bypass graft or coronary artery stent (Cardiac disorders) | 2 (2)
Significant structural heart disease (Cardiac disorders) | 1 (1)
Positive electrophysiology study findings (Cardiac disorders) | 1 (1)
Initiation of antiarrhythmia medical therapy (Cardiac disorders) | 2 (2)
Major adverse cardiac events [MACE] (Cardiac disorders) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-04-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT02683174/Prot_000.pdf